CLINICAL TRIAL: NCT04963478
Title: Study on Exercise Safety of Patients With Cardiovascular Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00006761-M2020073
Record Dates: First submitted 2021-06-27; First posted 2021-07-15 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-06

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Exercise

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: exercise — exercise testing

SUMMARY:
To retrospectively observe the cardiovascular safety during exercise in patients with cardiovascular diseases

ELIGIBILITY:
Inclusion Criteria:

Patients with confirmed or suspected cardiovascular disease who completed the trial

Exclusion Criteria:

Refusing to participate in the study

Ages: 19 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed or suspected cardiovascular disease who completed the trial from January 2008 to September 2019 at Peking University Third Hospital with complete data
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-08-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
exercise-related cardiovascular events | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Wei Zhao, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No